CLINICAL TRIAL: NCT04559425
Title: Slow Heart Registry: A Prospective Observational Cohort Study of Fetal Immune-mediated High Degree Heart Block
Brief Title: Slow Heart Registry of Fetal Immune-mediated High Degree Heart Block
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Edgar Jaeggi, Senior Associate Scientist Emeritus, The Hospital for Sick Children
Other Study IDs: 1000065121
Record Dates: First submitted 2020-09-11; First posted 2020-09-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Heart Block Complete; Heart Block Second Degree
Keywords: fetal; heart block; anti-Ro antibodies; steroids; outcome
MeSH Terms: conditions — Heart Block | interventions — Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective observational cohort 1: Complete AVB (3rd degree) diagnosed ≤ 32+0 weeks with or without hydrops
  Interventions: Drug: Dexamethasone; Other: No Dexamethasone
- Prospective observational cohort 2: Incomplete AVB (2nd; 2:1; 2nd-3rd degree) diagnosed ≤ 32+0 weeks with or without hydrops
  Interventions: Drug: Dexamethasone; Other: No Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — All management decisions are made by the primary physician and may include: 1) no treatment with dexamethasone or 2) treatment with dexamethasone from the time of enrollment
Other: No Dexamethasone — All management decisions are made by the primary physician and may include: 1) no treatment with dexamethasone or 2) treatment with dexamethasone from the time of enrollment

SUMMARY:
Few studies are specifically designed to address health concerns that are already relevant during pregnancy. The consequence is a lack of evidence on best clinical practice. This includes mothers and their babies when pregnancy is complicated by an abnormally slow heart rate due to maternal antibody-mediated heart disease in the unborn baby (fetus). Since the late seventies, it has been possible to detect and monitor fetal disease by ultrasound images and to treat selected conditions with pharmaceuticals administered via the mother. To this day, physicians need to make decisions about the management of such pregnancies without evidence from prospective clinical trials on drug efficacy and safety. The SLOW HEART REGISTRY is a multi-centered prospective observational study that will address the knowledge gap to guide future management of high-degree immune-mediated heart block to the best of care. The study seeks to establish an international database of the management and outcome of affected fetuses, to be used to publish information on the results of currently available prenatal care and to evaluate the need for additional research.

DETAILED DESCRIPTION:
The SLOW HEART REGISTRY is a multi-centered prospective observational study of fetuses diagnosed with high-degree immune-mediated atrio-ventricular heart block (AVB). The study seeks to establish an international database of the management and outcome of affected fetuses, to be used to publish information on the results of currently available prenatal care and to evaluate the need for additional research.

The study aims are to document the outcome of patients diagnosed prenatally with immune-mediated 2nd or 3rd degree AVB irrespective of the primary choice of prenatal care.

The primary objective will be to determine the rate of transplant-free survival to 1 year of life of fetuses with AVB based on the prenatal management decision:

* Cohort 1: Fetuses not treated with fluorinated glucocorticoids
* Cohort 2: Fetuses treated with fluorinated glucocorticoids from the time of immune-mediated AVB diagnosis.

Secondary objectives will be to determine:

1. the evolution of clinical findings from AVB diagnosis to birth (AV conduction; fetal heart rate; other NL manifestations; fetal growth; effusions/hydrops) between cohorts;
2. the need of new/additional treatment (steroids; beta-mimetics; IVIG) to birth;
3. gestational age and weight at birth;
4. postnatal management (pacing; steroids; IVIG); and
5. clinical evolution from birth to 1-3 years of life (cardiac function; developmental milestones; infant growth; health).

Prevalence of relevant fetal-maternal events and complications (death; IUGR; morbidity) between the study cohorts will also be determined.

All management is decided by the treating center and physicians in accordance to institutional guidelines and clinical findings. Patient enrollment in the SLOW HEART REGISTRY is possible within up to 8 days of the initial management decision.

Participation in this prospective observational cohort study requires site REB approval and an executed legal contract with the primary investigator/SickKids Hospital, Toronto.

ELIGIBILITY:
Inclusion Criteria:

* Written informed maternal consent to participate in the Slow Heart Registry
* High-degree (2nd; 2:1; 2nd-3rd or 3rd degree) AVB diagnosed ≤ 32+0 weeks with or without hydrops
* Enrollment within maximally 8 days of high-degree AVB diagnosis
* Positive or pending anti-Ro/La antibody test results at the time of enrollment

Exclusion Criteria:

* AVB associated with major CHD (e.g. left atrial isomerism, cc-TGA)
* AVB with known negative anti-Ro and/or La antibody test result at enrollment
* 1st degree AVB
* Sinus bradycardia with normal 1:1 AV conduction
* Blocked atrial bigeminy (irregular atrial rate with failure of AV conduction of the premature atrial beat)
* Primary delivery for postnatal treatment
* Maternal-fetal conditions (other than cardiac NL) associated with high odds of premature delivery or death (e.g. renal failure, significant infectious diseases, major extracardiac anomalies, PROM, etc.)
* Preexisting maternal mental disorder (e.g. bipolar, mania, severe depression, substance abuse)
* Poorly controlled insulin-dependent diabetes (HbA1c >7%) at CAVB diagnosis
* Oligohydramnios (deepest/maximal vertical pocket <2 cm)
* Severe IUGR (estimated fetal weight <3rd percentile)

Ages: 16 Years to 50 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Enrollment into the SLOW HEART Registry is possible within maximally 8 days of the fetal heart block diagnosis and a management decision to treat or not to treat. If a mother elects participation in the Registry, her treating physician will continue to provide care in accordance with clinical practice at the site and will decide all therapy including close observation without or with immediate steroid treatment.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from cardiac death ≥1 year of life | up to 12 months

SECONDARY OUTCOMES:
Proportion of participants with fetal and neonatal death and their causes/factors | 1 month
Proportion of participants with change in prenatal treatment | up to 6 months
Proportion of secondarily treated patients (initially untreated group 1 cases) | up to 6 months
Proportion of serious pregnancy outcomes (IUFD, IUGR <3rd percentile, delivery <35 weeks) | up to 6 months
Proportion of patients/group with progression from incomplete to complete AVB by 1 year | Fetal diagnosis to 12 months
Proportion of maternal serious adverse events and outcomes | Fetal diagnosis to 12 months
Average gestational age at birth | Birth
Average birth weight | Birth
Freedom from permanent pacemaker implantation from birth to 1 year of life | Birth to 12 months
Prevalence of significant heart failure (HF score, echo, HF treatment) at 1 year of life | 12 months
Proportion of children with moderate/severe neuro-developmental delay at 12-18 months | 12-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Jaeggi, MD, Principal Investigator — The Hospital for Sick Children, Toronto
Locations (27):
- United States (12):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Mercy Kansas City, Kansas City, Kansas
  - Boston Children's Hospital, Boston, Massachusetts
  - The Children's Heart Clinic/Children's Minnesota, Minneapolis, Minnesota
  - Columbia University (New York), New York, New York
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- National Heart Hospital, Sofia, Bulgaria
- Canada (2):
  - IWK Nova Scotia Health, Halifax, Nova Scotia
  - The Hospital for Sick Children, Toronto
- Hospital District of Helsinki and Uusimaa, Helsinki, Finland
- Grenoble University Hospital, Grenoble, France
- University of Bonn, Bonn, Germany
- Hong Kong Children's Hospital, Ngau Tau Kok, Hong Kong
- Japan (2):
  - Kanagawa Children's Medical Center, Kanagawa
  - Shizuoka Children's Hospital, Shizuoka
- Leiden University Medical Center - LUMC, Leiden, Netherlands
- Centre of Postgraduate Medical Education Poland, Warsaw, Poland
- Sweden (3):
  - Queen Silvia Children's Hospital, Gothenburg
  - Skane University Hospital in Lund, Lund
  - Karolinska University Hospital, Astrid Lindgen Childrens Hospital, Solna
- Taiji Clinic, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No